CLINICAL TRIAL: NCT05061303
Title: The Importance of the Use of Omeprazole and Famotidine in the Development of Chronic Dysfunction of the Transplanted Kidney
Brief Title: Omeprazole and Famotidine in Chronic Dysfunction of the Transplanted Kidney
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Miłosz Miedziaszczyk, Principal Investigator, Poznan University of Medical Sciences
Other Study IDs: 687/20
Record Dates: First submitted 2021-09-13; First posted 2021-09-29 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Kidney Rejection Transplant
Keywords: chronic kidney rejection process; tacrolimus; omeprazole; famotidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood samples

GROUPS / COHORTS (2):
- Group Omperazole: Patients will receive p.o. the standard, most commonly used triple immunosuppression regimen: tacrolimus, mycophenolate mofetil, prednisone and p.o. omeprazole 20 mg (group Omeprazole).
  Interventions: Other: Assessment of the drug concentration in the blood
- Group Famotidine: Patients will receive p.o. the standard, most commonly used triple immunosuppression regimen: tacrolimus, mycophenolate mofetil, prednisone and p.o. famotidine 20 mg (group Famotidine).
  Interventions: Other: Assessment of the drug concentration in the blood

INTERVENTIONS:
Other: Assessment of the drug concentration in the blood — The material in the study will be blood, in which tacrolimus concentrations will be measured at the following time points: 0, 2hours, 6hours, 12hours after drug administration, without taking omeprazole/famotidine and then the next day after taking the protective drug in same time points, without 12hours. Sequentially routinely in the so-called point T0 before taking the drug (12 hours after the last dose) during follow-up visits at the Transplant Outpatient Clinic.

SUMMARY:
The aim of the study is to compare the effect of omeprazole and famotidine on the risk of developing chronic renal transplant dysfunction. For the study, it is planned to qualify 24 stabilized adult patients from 1-24 months after kidney transplantation, who will receive p.o. the standard, most commonly used triple immunosuppression regimen: tacrolimus, mycophenolate mofetil, prednisone and depending on the group p.o.: omeprazole 20 mg (group I) or famotidine 20 mg (group II). The material in the study will be blood, in which tacrolimus concentrations will be measured at the following time points: 0, 2h, 6h, 12h after drug administration, without taking omeprazole/famotidine and then the next day after taking the protective drug in same time points, without 12h. Sequentially routinely in the so-called point T0 before taking the drug (12 hours after the last dose) during follow-up visits at the Transplant Outpatient Clinic. Tacrolimus concentrations will be determined using the Chemiluminescent Microparticle Immuno Assay method. As standard, laboratory tests will be performed during follow-up visits.

In addition, it is planned to assess titer of donor-specific antibodies at the time of qualification and then after 18 months, immunological profile (flow cytometry) at the time of qualification and then after 18 months, and concentration in serum and urine of a potential marker of progression and decrease in glomerular filtration - kidney injury molecule-1 at the time of qualification and then after 18 months. The obtained results will be correlated with the histopathological evaluation of the transplanted kidney in the case of organ biopsy performed on clinical indications.

Comparative statistical analysis of drug concentration values will be carried out. Additionally, genetic tests will be performed to assess the patient's metabolic variant for CYP2C19. Due to the potential influence of omeprazole on the pharmacokinetics of tacrolimus, which may influence the process of chronic rejection of the transplanted kidney and drug toxicity, it seems important to study this hypothesis, as well as researching for therapeutic substances neutral to the above process. The use of famotidine in place of omeprazole may turn out more beneficial and safer for renal transplant patients. During follow-up visits at the Transplant Clinic at the Department and Clinic of Nephrology, Transplantology and Internal Diseases, changes in blood concentrations of tacrolimus are noticed. Related reasons are being looked for. The above study will confirm or reject the relationship of changes in tacrolimus levels with omeprazole. It is planned to present the results at a scientific conference. The research results will be published in a scientific journal.

DETAILED DESCRIPTION:
1. Scientific aim of the project Tacrolimus is an immunosuppressive calcineurin inhibitor used to prevent rejection in allogeneic organ transplant recipients such as kidney, liver, heart or lungs. It is metabolized in the liver with the participation of the cytochrome P450 isoform CYP3A4 (CYP3A4), it is characterized by a narrow therapeutic window, dose-dependent toxicity and high inter-individual and intra-individual variability. Increased serum concentration of tacrolimus may be caused by substrates and inhibitors of CYP3A4, revealing adverse effects of this drug, especially nephrotoxicity. Proton pump inhibitors (PPIs) are used as standard in kidney transplant patients to prevent duodenal and gastric ulcer disease in connection with the use of glucocorticoids. One of the PPIs is omeprazole, which is a substrate and inhibitor of the enzyme CYP2C19 and CYP3A4 and also an inhibitor of P-glycoprotein. The enzyme CYP2C19 is mainly responsible for the metabolism of omeprazole, however, upon saturation or in the event of a mutation in the CYP2C19 gene (a poor metabolizer), CYP3A4 becomes the major enzyme involved in the elimination of omeprazole and thus may interact with tacrolimus. Therefore, it seems important to use drugs with a similar prophylactic effect on the gastrointestinal tract, which, unlike omeprazole, are not substrates or inhibitors of the CYP3A4 enzyme, such as famotidine - an antagonist of H2 receptors.

   Due to the potential influence of omeprazole on the pharmacokinetics of tacrolimus, which may influence the process of chronic rejection of the transplanted kidney and drug toxicity, it seems important to study this hypothesis, as well as researching for therapeutic substances neutral to the above process. The use of famotidine in place of omeprazole may turn out more beneficial and safer for renal transplant patients. The aim of the study is to compare the effect of omeprazole and famotidine on the risk of developing chronic renal transplant dysfunction.
2. Project meaning No study has been found in the available scientific literature to assess the effect of omeprazole administration on the development of chronic renal transplant rejection. However, studies have been found to assess the effect of omeprazole on the change in tacrolimus plasma levels. The search strategy consisted of controlled vocabulary and keywords. The following databases were searched: MEDLINE (Pubmed), Scopus, Web of Science and Cochrane. The main search concept was to combine "tacrolimus", "omeprazole" and "kidney". 74 studies were found, of which only 7 were related to the topic searched.

   In one of the studies, the authors presented a case of a patient and observed a change in the concentration of tacrolimus in the blood plasma after switching from ranitidine to omeprazole. Since informed consent could not be obtained from this patient, authors were unable to access the genetic information. It was not known if the patient had a mutation in the gene encoding CYP2C19. Other authors observed an over fourfold increase in the concentration of tacrolimus after the administration of omeprazole. Patient was homozygous mutated (*2/*2) for CYP2C19, carrying an aberrant splicing site that reduces significantly or inactivates the encoded protein's activity of CYP2C19, classified as CYP2C19 poor metabolizer. The CYP2C19 gene, which includes nine exons and eight introns, is located at the 10q24.1-10q24.3 locus of chromosome 10, where coding sequences is 1,473 bp and resulting in a protein of 490 amino acid residues. Approximately 25 genetic variants in the exonic region of the CYP2C19 have been identified. CYP2C19 is involved in metabolizing several important therapeutic drugs, including omeprazole. Common variants of the CYP2C19 gene are associated with impaired drug metabolism. CYP2C19*2 and CYP2C19*3 were identified in individuals who exhibited a reduced capability for metabolizing the probe drugs, and variant CYP2C19*17 is associated with ultra-rapid metabolism of CYP2C19 substrates. The principal detrimental allele, CYP2C19*2, results from a guanine (G) to adenine (A) transition at position 681 in exon 5 (rs4244285), producing an aberrant splice site and it represents the most frequent CYP2C19 defect in all populations. CYP2C19*2 and CYP2C19*3 are the most common alleles, encoding enzymes with decreased activity. CYP2C19*3 (636G>A) is considered the most important allele, in which a point mutation in exon 4 results in a premature stop codon, and therefore nonfunctional protein. The prevalence of the CYP2C19 poor metabolizer (PM) phenotype is 2-5% among Caucasians and Africans, and ~15% in Asians, while CYP2C19*3 is considered to be an Asian mutation. CYP2C19*2 and *3 alleles have been proposed to explain <50%, to >90%, of the PM phenotype. The enzyme CYP2C19 is mainly responsible for the metabolism of omeprazole, however, in the event of a mutation in the CYP2C19 gene (poor metaboliser), CYP3A4 becomes the major enzyme involved in the elimination of omeprazole. Tacrolimus is also metabolised by CYP3A4, so in the above situation there is a competitive competition for the CYP3A4 enzyme, as a result, the metabolism of tacrolimus may be insufficient, and this may result in an increase in plasma tacrolimus concentrations, which may be a factor in the process of chronic renal rejection. In one of the studies, the authors demonstrated during study of 75 patients that recipients with CYP2C19*2/*2 genotype showed allograft delayed function (acute tubular necrosis in 3 patients) during treating with tacrolimus and omeprazole. It should be noted that other authors in clinical-analytical study (n = 51) conclused that an omeprazole- tacrolimus interaction is not clinically relevant. Despite possible competition or interaction at the molecular level, clinical management was not significantly affected in renal allograft recipients. However, the study lasted 6 months. The duration of the study was too short to provide an answer regarding the effect of tacrolimus on chronic renal rejection. In one of the works, the authors suggest in their study (n=27) that omeprazole may increase the serum tacrolimus concentration if ingested 2 hr before tacrolimus ingestion, likely through alkalization of the intestinal contents. Famotidine does not interact with the cytochrome P450-linked drug metabolizing enzyme system, therefore it is a good candidate for use in place of omeprazole.

   It is known that there may be an interaction between omeprazole and tacrolimus. There have been several cases of such an interaction in history. It is not known whether the use of omeprazole has an impact on the chronic rejection of a transplanted kidney. The scheduled study is a new issue. Conducting the above study will allow to assess whether the use of omeprazole has an impact on the process of chronic rejection of the transplanted kidney.

   Due to the timing of kidney rejection, there are three phases: hyperacute, acute and chronic phase. Hyperacute rejection occurs immediately after transplantation and is associated with the presence in the blood of the recipient of antibodies that react with antigens on the organ donor endothelial cells. They are mainly antibodies against HLA antigens and against AB0 blood group antigens. Acute rejection occurs within a few days to several months after transplantation. It can be cellular, humoral or mixed. Cellular response mechanisms (cellular rejection) dominate the pathogenesis of acute rejection. Chronic rejection occurs one year after transplantation. Due to the type of reaction, it may be cellular, humoral or mixed with a predominance of cellular or antibody-dependent mechanisms. To the current knowledge, donor-specific antibodies are mainly responsible for late graft loss.

   With the introduction of tissue typing tests, antibody-mediated hyperacute rejection of the kidney is rarely observed. With the immunosuppression currently available, acute T-cell mediated rejection has become a rare event. In contrast, chronic antibody-mediated rejection is considered to be a major contributor to graft loss in the late posttransplant phase. Today there is still noeffective strategy to treat this indolent and slowly progressing form of antibody-mediated rejection. Therefore, the aim of our study focuses on the chronic rejection of a transplanted kidney.

   In the available scientific literature (MEDLINE (Pubmed), Scopus, Web of Science and Cochrane) no study was found to assess the effect of omeprazole and famotidine in the development of chronic renal transplant dysfunction. During follow-up visits at the Transplant Clinic at the Department and Clinic of Nephrology, Transplantology and Internal Diseases, changes in blood concentrations of tacrolimus are noticed. Related reasons are being looked for. The above study will confirm or reject the relationship of changes in tacrolimus levels with omeprazole.

   It is anticipated that the co-administration of omeprazole and tacrolimus will be more difficult to keep tacrolimus levels within the therapeutic range than in the combination of famotidine with tacrolimus. As a result, drug interaction may be one of the risk factors for the development of chronic renal transplant dysfunction, and the use of famotidine instead of omeprazole may prove to be more beneficial and safer for renal transplant patients. The study may change the current immunosuppression regimen that is used around the world. It is planned to present the results at a scientific conference. The research results will be published in a scientific journal. The research will be the basis for publications, and these, as a series of publications, will form the basis of the doctoral dissertation.

   Alternative hypothesis In a situation where I did not achieve statistical significance between the groups, I planned to test the genotype of patients who would show the greatest deviations in the concentration of tacrolimus in the blood plasma in the group receiving omeprazole. This will confirm the relationship of the mutations in the CYP2C19 gene with changes in tacrolimus concentration.

   Access to research equipment The Clinical Hospital of Heliodor Święcicki has laboratory diagnostics and the method of tacrolimus determination used in the project. The kidney injury molecule - 1 marker will also be tested at the hospital. The Chair and Department of Nephrology, Transplantology and Internal Diseases collaborates with the immunology laboratory (Chair of Clinical Immunology of Poznan University of Medical Sciences) where the immune profile tests will be performed. Genetic tests will be performed by an external company (outsourcing). The titre of donor specific antibodies will be performed at the HLA Tissue Compatibility Laboratory with the Laboratory of Genetic Diagnostics (Regional Center for Blood Donation and Haemotherapy in Poznań).
3. Research methodology For the study, it is planned to qualify stabilized adult patients from 1-24 months after kidney transplantation. The group size was estimated at 36, taking into account the size of the kidney transplant population (550,000), estimates that the studied trait was found in 10% of the population, the confidence level was set at 95%, and the maximum error at 10%. On the day of enrollment in the study, the following data will be collected: age, sex, weight, height, BMI, living donor / dead donor, cold ischemia time, delayed graft function (hemodialysis), acute rejection process, comorbidities (diabetes, hypertension), CMV. Tacrolimus concentrations will be determined using the Chemiluminescent Microparticle Immuno Assay method (CMIA) - instrument Alininity i. As standard, laboratory tests (creatinine, eGFR, urinalysis, urinalysis, hemoglobin, leukocytes, neutrophils, proteinuria, CRP) will be performed during follow-up visits. In addition, it is planned to assess titer of donor-specific antibodies (solid-phase assay as HLA antigen-coated bead method [Luminex] - instrument Luminex) at the time of qualification and then after 18 months, immunological profile (flow cytometry method - instrument Facscalibur) at the time of qualification and then after 18 months and concentration in serum and urine of a potential marker of progression and decrease in glomerular filtration - kidney injury molecule-1 at the time of qualification and then after 18 months (colorimetric method - instrument Colorimeter). The obtained results will be correlated with the histopathological evaluation of the transplanted kidney in the case of organ biopsy performed on clinical indications. In the final stage, a comparative statistical analysis of drug concentration values and other statistical tests will be carried out. The student's T-test will check if there is a normal distribution. The Fisher- Snedecor test will assess whether the variances in populations are equal or different. Then the Student T-test for independent groups or the Student T-test with Cochran-Cox correction will be applied. Additionally, genetic tests will be performed to assess the patient's metabolic variant for CYP2C19. For cost reasons, these studies will be performed only for patients who will show significant changes in tacrolimus concentrations.

ELIGIBILITY:
Inclusion Criteria:

* receiving of p.o. the standard, most commonly used triple immunosuppression regimen: tacrolimus, mycophenolate mofetil, prednisone and omeprazole or famotidine,
* stabilized adult patients from 1-24 months after kidney transplantation

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the study, it is planned to qualify stabilized adult patients from 1-24 months after kidney transplantation, who will receive p.o. the standard, most commonly used triple immunosuppression regimen: tacrolimus, mycophenolate mofetil, prednisone and omeprazole 20 mg or famotidine 20 mg.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-10-17 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the drug concentration in the blood | Sequentially routinely in the so-called point T0 before taking the drug (12 hours after the last dose) during follow-up visits at the Transplant Outpatient Clinic.
  The material in the study will be blood, in which tacrolimus concentrations will be measured at the following time points: 0, 2h, 6h, 12h after drug administration, without taking omeprazole/famotidine and then the next day after taking the protective drug in same time points, without 12h. Sequentially routinely in the so-called point T0 before taking the drug (12 hours after the last dose) during follow-up visits at the Transplant Outpatient Clinic.
Change from Baseline titer of donor-specific antibodies | 0, 6, 12, 18 Month
  Change from Baseline donor-specific antibodies after 18 months.
Change from Baseline immunological profile (flow cytometry) - Th2 to Th1 ratio | 0, 18 Month
  Change from Baseline immunological profile (flow cytometry) - Th2 to Th1 ratio after 18 months.
Change from Baseline concentration in serum and urine of a potential marker of progression and decrease in glomerular filtration - kidney injury molecule-. | 0, 18 Month
  Change from Baseline concentration in serum and urine of a potential marker of progression and decrease in glomerular filtration - kidney injury molecule-1 after 9 and 18 months.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Hospital in Poznan of the Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takahashi K, Yano I, Fukuhara Y, Katsura T, Takahashi T, Ito N, Yamamoto S, Ogawa O, Inui K. Distinct effects of omeprazole and rabeprazole on the tacrolimus blood concentration in a kidney transplant recipient. Drug Metab Pharmacokinet. 2007 Dec;22(6):441-4. doi: 10.2133/dmpk.22.441. PMID 18159131
- [Background] Moreau C, Debray D, Loriot MA, Taburet AM, Furlan V. Interaction between tacrolimus and omeprazole in a pediatric liver transplant recipient. Transplantation. 2006 Feb 15;81(3):487-8. doi: 10.1097/01.tp.0000194861.59543.b9. No abstract available. PMID 16477241
- [Background] Zhao W, Fakhoury M, Maisin A, Baudouin V, Storme T, Deschenes G, Jacqz-Aigrain E. Pharmacogenetic determinant of the drug interaction between tacrolimus and omeprazole. Ther Drug Monit. 2012 Dec;34(6):739-41. doi: 10.1097/FTD.0b013e318271b6e6. PMID 23042259
- [Background] Hosohata K, Masuda S, Katsura T, Takada Y, Kaido T, Ogura Y, Oike F, Egawa H, Uemoto S, Inui K. Impact of intestinal CYP2C19 genotypes on the interaction between tacrolimus and omeprazole, but not lansoprazole, in adult living-donor liver transplant patients. Drug Metab Dispos. 2009 Apr;37(4):821-6. doi: 10.1124/dmd.108.025833. Epub 2009 Jan 12. PMID 19139162
- [Background] Maguire M, Franz T, Hains DS. A clinically significant interaction between tacrolimus and multiple proton pump inhibitors in a kidney transplant recipient. Pediatr Transplant. 2012 Sep;16(6):E217-20. doi: 10.1111/j.1399-3046.2011.01559.x. Epub 2011 Aug 23. PMID 21883747
- [Background] Boso V, Herrero MJ, Bea S, Galiana M, Marrero P, Marques MR, Hernandez J, Sanchez-Plumed J, Poveda JL, Alino SF. Increased hospital stay and allograft dysfunction in renal transplant recipients with Cyp2c19 AA variant in SNP rs4244285. Drug Metab Dispos. 2013 Feb;41(2):480-7. doi: 10.1124/dmd.112.047977. Epub 2012 Nov 21. PMID 23175667
- [Background] Pascual J, Marcen R, Orea OE, Navarro M, Alarcon MC, Ocana J, Villafruela JJ, Burgos FJ, Ortuno J. Interaction between omeprazole and tacrolimus in renal allograft recipients: a clinical-analytical study. Transplant Proc. 2005 Nov;37(9):3752-3. doi: 10.1016/j.transproceed.2005.09.126. PMID 16386527
- [Background] Peloso LJ, Faria PN, Bossolani MV, de Oliveira HB, Ferreira Filho SR. The serum concentration of tacrolimus after ingesting omeprazole: a pilot study. Transplantation. 2014 Sep 27;98(6):e63-4. doi: 10.1097/TP.0000000000000351. No abstract available. PMID 25221905
- [Background] Mei S, Wang J, Chen D, Zhu L, Zhao M, Tian X, Hu X, Zhao Z. Simultaneous determination of cyclosporine and tacrolimus in human whole blood by ultra-high performance liquid chromatography tandem mass spectrometry and comparison with a chemiluminescence microparticle immunoassay. J Chromatogr B Analyt Technol Biomed Life Sci. 2018 Jun 15;1087-1088:36-42. doi: 10.1016/j.jchromb.2018.04.028. Epub 2018 Apr 13. PMID 29704799
- [Background] Shahbaz SK, Pourrezagholi F, Barabadi M, Foroughi F, Hosseinzadeh M, Ahmadpoor P, Nafar M, Yekaninejad MS, Amirzargar A. High expression of TIM-3 and KIM-1 in blood and urine of renal allograft rejection patients. Transpl Immunol. 2017 Aug;43-44:11-20. doi: 10.1016/j.trim.2017.07.002. Epub 2017 Jul 27. PMID 28757398
- [Derived] Miedziaszczyk M, Karczewski M, Idasiak-Piechocka I. The effect of the use of omeprazole versus famotidine on the kidney transplant function: a randomized controlled study. Sci Rep. 2025 Jan 13;15(1):1805. doi: 10.1038/s41598-025-85534-w. PMID 39805983
- [Derived] Miedziaszczyk M, Karczewski M, Grabowski T, Wolc A, Idasiak-Piechocka I. Assessment of omeprazole and famotidine effects on the pharmacokinetics of tacrolimus in patients following kidney transplant-randomized controlled trial. Front Pharmacol. 2024 Apr 4;15:1352323. doi: 10.3389/fphar.2024.1352323. eCollection 2024. PMID 38638867